CLINICAL TRIAL: NCT00754442
Title: Clinical and Molecular Characterization of Suspected Partial 25-hydroxyvitamin D-1-alpha-hydroxylase Deficiency
Brief Title: Suspected Deficient Activation of Vitamin D in Patients With Secondary Hyperparathyroidism
Acronym: 1hydroxylase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Elizabeth Streeten, Associate Professor of Medicine, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-28679; H-28679 (Other: IRB number)
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Results first posted 2014-05-14 (Estimated); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Secondary Hyperparathyroidism
Keywords: hyperparathyroidism; parathyroid; vitamin D; vitamin D deficiency
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Hyperparathyroidism; Vitamin D Deficiency | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- teriparatide control (Active Comparator): control subject
  Interventions: Drug: Teriparatide
- Teriparatide Patient (Experimental): Patient with secondary hyperparathyroidism
  Interventions: Drug: Teriparatide

INTERVENTIONS:
Drug: Teriparatide — Teriparatide will be given by continuous intravenous infusion at a rate of 12 pmol/kg/hr for 8 hours to both "patients" and "controls"
  Other Names: Forteo

SUMMARY:
The purpose of this study is to determine if a reduction in the enzyme 1-hydroxylase, which activates Vitamin D, is the cause of overactivity of the parathyroid glands (called secondary hyperparathyroidism - normal blood calcium and elevated parathyroid hormone) in a selected group of young patients with normal kidney function.

DETAILED DESCRIPTION:
Vitamin D, an essential nutrient, is produced by the skin after sunlight shines on it. Vitamin D must then be activated by both the liver and the kidneys to perform its function of maintaining strong bones and helping to prevent heart disease, infection, diabetes and cancer. Reduced kidney activation of Vitamin D occurs with advanced age and with all kidney diseases. We have identified a small group of patients who appear to have reduced ability of the kidneys to activate vitamin D, even though they are young and do not have chronic kidney disease. In these patients, we are comparing the ability of their kidneys to activate Vitamin D to that of healthy controls. To stimulate the kidneys to activate Vitamin D, we are giving parathyroid hormone intravenously over 8 hours and collecting blood and urine at baseline, 4 and 8 hours. This type of parathyroid infusion does not cause side effects. The gene that controls this activation is also being studied (by a simple blood test) to look for abnormalities. We are now actively recruiting healthy controls for this study.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian female
* Age 40-59 years
* Serum creatinine < 1.3 and estimated glomerular filtration rate (GRF) > 60
* Serum calcium in the normal range (for U Md lab 8.6-10 mg/dl)
* Parathyroid hormone in the normal range (for U Md lab 12-54 pg/ml)
* Normal 25-hydroxyvitamin D level (30 ng/ml or higher)
* For women of childbearing age, non-pregnant (based on negative urine pregnancy test on the morning of the teriparatide infusion)

Exclusion Criteria:

* Non-caucasian
* Age under 40 and over 59 years
* Male
* Serum creatinine over 1.3 or estimated glomerular filtration rate (GFR) < 60
* Abnormal serum calcium (for U Md lab, below 8.6 or above 10 mg/dl)
* Abnormal parathyroid hormone (for U Md lab, above 65 or below 12 pg/ml)
* For women of childbearing age, non-pregnant (based on urine pregnancy test on the morning of the teriparatide infusion)
* History of bone radiation
* History of Paget disease of bone
* History of bone malignancy or metastases
* History of allergy or sensitivity to Forteo

Ages: 40 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Streeten, MD, Principal Investigator — Division of Endocrinology, University of Maryland School of Medicine
Locations (1):
- University of Maryland School of Medicine Division of Endocrinology, Baltimore, Maryland, United States

REFERENCES:
- [Result] Streeten EA, Rogstad AS, Flammer KM, Zarbalian K, Ryan K, Horwitz M, Holick MF, Shelton J. Reduced parathyroid hormone-stimulated 1,25-dihydroxyvitamin d production in vitamin d sufficient postmenoposual women with low bone mass and idiopathic secondary hyperparathyroidism. Endocr Pract. 2013 Jan-Feb;19(1):91-9. doi: 10.4158/EP12151.OR. PMID 23186957

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All in the "patient" group were recruited from the Metabolic Bone Clinic at U Md, except one, who was recruited from prior participation in the Amish Family Osteoporosis Study, recruited from 3/15/07-11/14/08
Pre-assignment Details: Of 11 "controls" enrolled, 6 completed the study and 5 dropped out because they didn't want to do the parathyroid hormone (PTH) infusion. Of 9 "patients" recruited, 6 completed the study. The others were excluded after their screening labs showed that their renal function was below the inclusion criteria.
Groups:
- Controls: controls with normal PTH
- Patient Group: patients with secondary hyperparathyroidism
Period: Overall Study
Arm/Group | Controls | Patient Group
Started | 11 (controls 11) | 9 (patients 9)
Completed | 6 | 6
Not Completed | 5 | 3
Not completed — Withdrawal by Subject | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Controls | Patient Group | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (4.4) | 53.0 (2.5) | 52.4 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: The Level of Activated Vitamin D (1,25-dihydroxyvitamin D) After Parathyroid Hormone Infusion at Baseline, 4 and 8 Hours
Description: 1,25-D was measured at baseline, 4 and 8 hours after PTH infusion
Time Frame: baseline, 4 and 8 hours after start of infusion
Population: The final analysis was made on participants with glomerular filtration rate (GFR) of 70 and above since <70, 1,25-D production decreases. After study completion, it was noted that one participant in each group (patient and control) had GFR<70 so these two participants were excluded from final analysis.
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Group 1: "patients" with secondary hyperparathyroidism
- Controls: Controls without secondary hyperparathyroidism
Arm/Group | Group 1 | Controls
Number analyzed (Participants) | 5 | 5
pg/ml
  Baseline | 40.6 (5.6) | 46.2 (3.7)
  4 hours | 39.8 (6.0) | 58.8 (6.7)
  8 hours | 56.4 (9.2) | 105 (2.3)
Statistical Analysis 1: Comparison: Group 1 vs Controls; The null hypothesis is that there is no statistical difference between patients and controls at baseline; Test type: Superiority or Other; p = 0.1, t-test, 2 sided — see above; 95%
Statistical Analysis 2: Comparison: Group 1 vs Controls; The null hypothesis is that there is no statistical difference between patients and controls at 4 hours; Test type: Superiority or Other; p = 0.002, t-test, 2 sided
Statistical Analysis 3: Comparison: Group 1 vs Controls; The null hypothesis is that there is no statistical difference between patients and controls at 8 hrs; Test type: Superiority or Other; p = 0.003, t-test, 2 sided

2. Secondary Outcome: The Number of Patients With Mutations in CYP27B1
Description: CYP27B1 gene (the gene for 25-hydroxyvitamin D-1-alpha hydroxylase) was sequenced for all in patient group and compared with published control data
Time Frame: blood samples taken at baseline and sequenced over several days
Population: All patients were sequenced and compared to published control data. Controls were not sequenced for cost reasons
Measure: Number; unit: participants
Groups:
- Patients: patients with idiopathic secondary hyperparathyroidism
Arm/Group | Patients
Number analyzed (Participants) | 9
participants | 0 (5)

ADVERSE EVENTS:
Time Frame: During PTH infusion, 2 participants, one in patient and one in control groups had one episode of vomiting each.
Arm/Group | Controls | Patient Group
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 1/11 | 1/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Controls (N=11) | Patient Group (N=9)
vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) — One patient and one control each had one episode of vomiting during the PTH infusion. Both continued the full 8 hrs of infusion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No